CLINICAL TRIAL: NCT01497080
Title: Distal Radius Fracture Prospective Database 50-80 Years Old Overview: "Identification of Risk of Adverse Activity Transition Following a Distal Radius Fracture".
Brief Title: Distal Radius Fracture Prospective Database 50-80 Years Old
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Joy MacDermid, Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 18482
Record Dates: First submitted 2011-12-19; First posted 2011-12-22 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Radius Fracture Distal
Keywords: distal radius fracture; Condition; risk factors; adverse activity transitions following DRF; optimal assessment approach
MeSH Terms: conditions — Wrist Fractures; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1
- activity level
- no treatment

SUMMARY:
The Problem Distal radius fractures (DRF) are common and result in a variable amount of disability. The investigators have completed considerable work in developing tools that measure impairment and disability after DRF . The investigators initial studies indicate that the associated disablement process is multifactorial and variable with only 25% of the resultant disability predicted by baseline patient and injury characteristics. The investigators see DRF as a signal event where some people are at-risk of transitioning from an active lifestyle to inactivity and subsequent health risks. The investigators recent data confirms variable participation following a DRF. The traditional focus in orthopedic/rehabilitative approaches to DRF fracture management has been localized to the wrist, largely ignoring this potential transition and its health impacts. The investigators will initiate a line of investigation that will profile the at-risk older adult who presents with a DRF with the ultimate goal of accurate identification and prevention of adverse activity transitions (active to inactive). In this study the investigators will identify the extent of the problem by quantifying changes in activity/participation and its short-term health impacts. The investigators will also identify the risk factors present at time of injury that predict a loss of mobility/activity/participation. This work has the potential to identify tools and/or clinical prediction rules that identify at-risk individuals at a critical time where early intervention might most easily prevent adverse outcomes associated with inactivity.

ELIGIBILITY:
Inclusion Criteria:

individuals 50-80 years old

* one month of fracture resulting from a fall from standing height or less will be recruited through our orthopedic surgeon
* wrist fracture

Exclusion Criteria:

previous history of humeral, hip or vertebral fracture

• Testing will not be performed on patients with evident postural instability, severe chronic conditions (Parkinson's disease) or other vestibulo-ocular abnormalities.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants aged 50-80 years of age who have incurred a wrist fracture
Sampling Method: Probability Sample
Enrollment: 195 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joy MacDernmid, PhD, Principal Investigator — St. Joseph's Health Care London
Locations (1):
- HULC, St Joseph's health Care London, London, Ontario, Canada

REFERENCES:
- [Background] Colquhoun HL, Letts LJ, Law MC, MacDermid JC, Missiuna CA. A scoping review of the use of theory in studies of knowledge translation. Can J Occup Ther. 2010 Dec;77(5):270-9. doi: 10.2182/cjot.2010.77.5.3. PMID 21268509
- [Background] Grewal R, MacDermid JC, Pope J, Chesworth BM. Baseline predictors of pain and disability one year following extra-articular distal radius fractures. Hand (N Y). 2007 Sep;2(3):104-11. doi: 10.1007/s11552-007-9030-x. Epub 2007 Mar 23. PMID 18780068